CLINICAL TRIAL: NCT01147107
Title: Hepatic Safety of Raltegravir-based and Efavirenz-based Antiretroviral Regimens in Antiretroviral-Naïve HIV-infected Subjects Co-Infected With Hepatitis C
Brief Title: Hepatic Safety of Raltegravir Versus Efavirenz as HIV Therapy for Patients With HIV and HCV Coinfection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Viet Tiep Hospital (Other); Oxford University Clinical Research Unit, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHARP 001
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C, Chronic; HIV Infection
Keywords: HIV/HCV co-infection; Antiretroviral therapy
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir based therapy (Experimental): Emtricitabine/tenofovir DF* 200 mg/300 mg po daily + Raltegravir 400 mg twice daily
  Interventions: Drug: Raltegravir
- Efavirenz based therapy (Active Comparator): Emtricitabine/tenofovir DF* 200 mg/300 mg po daily + Efavirenz 600 mg po daily
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Raltegravir — Emtricitabine/tenofovir DF* 200 mg/300 mg po daily + Raltegravir 400 mg twice daily
  Other Names: Isentress
  Arms: Raltegravir based therapy
Drug: Efavirenz — Emtricitabine/tenofovir DF* 200 mg/300 mg po daily + Efavirenz 600 mg po daily
  Other Names: Sustiva
  Arms: Efavirenz based therapy

SUMMARY:
The main objective is to evaluate the hepatic safety of raltegravir when compared to efavirenz, both in combination with tenofovir and emtricitabine as first-line HIV treatment in patients with HIV and hepatitis C coinfection.

DETAILED DESCRIPTION:
The trial will recruit 80 treatment-naive HIV-infected patients with chronic hepatitis C coinfection from two HIV treatment centers in Vietnam. Patients will be randomized to receive either raltegravir or efavirenz, both in combination of tenofovir and emtricitabine, as first-line HIV therapy over a period of 72 weeks. The primary endpoint is the rate of alanine aminotransferase (ALT) elevation during the 72 week study period. Secondary endpoints include rates of virological suppression, CD4 count change, numbers of AIDS events and death, rates of fasting glucose and cholesterol measures, neurocognitive function and levels of immune activation. Patients will be followed monthly for the first 3 months and every 3 months thereafter. At the end of the trial period, patients will be transferred to the National HIV treatment program for continuation of HIV therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients, age >18 years, meet Vietnam guideline to begin ART (CD4 count < 350 cells/mm3 and/or WHO stage III or IV disease)
* Hepatitis C infection as documented by positive HCV antibodies and a detectable serum HCV RNA level
* AST and ALT ≤ 2 x ULN (≤ 80 U/L)
* Estimated creatinine clearance ≥ 60 mL/min

Exclusion Criteria:

* Any prior ART
* Positive Hepatitis B surface antigen
* Clinical evidence of de-compensated cirrhosis (ascites, encephalopathy, esophageal bleeding)
* Requirement for acute therapy for other AIDS-defining illness within 14 days prior to study entry
* Currently on rifampicin therapy
* In the first trimester of pregnancy, intent to become pregnant, or breast feeding during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Van Vinh Chau Nguyen, MD, PhD, Principal Investigator — Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam; Cecilia M Shikuma, M.D., Principal Investigator — University of Hawaii - Hawaii Center for AIDS (HICFA); Thuy Le, M.D., Study Director — University of Hawaii, Oxford University Clinical Research Unit
Locations (2):
- Vietnam (2):
  - Viet Tiep General Hospital, Haiphong
  - Hospital for Tropical Diseases, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers upon request following the publication of the data. Researchers will contact the PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raltegravir Based Therapy | Efavirenz Based Therapy
Started | 39 | 41
Completed | 33 | 40
Not Completed | 6 | 1
Not completed — Lack of Efficacy | 5 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Based Therapy | Efavirenz Based Therapy | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Median (Full Range); unit: years] | 32 [31 to 34] | 33 [31 to 35] | 32 [31 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 32 | 37 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 41 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Rates of Grade 2 and Higher Alanine Aminotransferase (ALT) Elevations
Description: To estimate the rates of grade 2*and higher ALT elevations in the two regimens.
Time Frame: over week 72
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir Based Therapy | Efavirenz Based Therapy
Number analyzed (Participants) | 38 | 41
Participants | 24 | 30

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | Raltegravir Based Therapy | Efavirenz Based Therapy
All-Cause Mortality (participants affected / at risk) | 2/38 | 3/41
Serious Adverse Events (participants affected / at risk) | 8/38 | 8/41
Other Adverse Events (participants affected / at risk) | 21/38 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir Based Therapy (N=38) | Efavirenz Based Therapy (N=41)
Car Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicide (General disorders) | 0 (0) | 1 (1)
Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Infectious Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
CNS Syndrome Unclear Etiology (Nervous system disorders) | 0 (0) | 1 (1)
PCP Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bacterial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PML (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir Based Therapy (N=38) | Efavirenz Based Therapy (N=41)
ALT Elevation (Hepatobiliary disorders) | 21 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No